CLINICAL TRIAL: NCT01282125
Title: A Comparative Study of Nasal Obstruction in a Sleep Apnea Population Compared to the General Population
Brief Title: Nasal Obstruction in Sleep Apnea Patients Compared to the General Population
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Sorlandet Hospital HF (Other Government)
Responsible Party: Sponsor
Other Study IDs: OSAS og nasalstenose
Record Dates: First submitted 2011-01-18; First posted 2011-01-24 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Obstructive Sleep Apnoea Syndrome; Nasal Obstruction
Keywords: general population; prevalence; Norway
MeSH Terms: conditions — Sleep Apnea, Obstructive; Nasal Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- sleep apnea: 100 patients suffering from obstructive sleep apnea syndrome
- controls: 100 subjects matching cases to age, sex, and body weight

SUMMARY:
Recent clinical findings of research at Trondheim University Hospital suggest that surgical correction of the nose septum in addition to volume reduction of the nose cavity may be beneficial in patients who suffer from both nose obstruction and obstructive sleep apnea syndrome(data not yet published).

This study aims to compare nose obstruction prevalence in sleep apnea patients and the general population

ELIGIBILITY:
Inclusion Criteria:

* ???

Exclusion Criteria:

* ???

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients: St Olavs Hospital, Trondheim, Norway Controls: Community sample, residents of Trøndelag, Norway
Sampling Method: Non-Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
patient reported nasal obstruction | 1 week
  assessed by a 10-point visual analogue scale (VAS) and Sino Nasal Outcome Score(SNOT-20) questionnaire.
objective nasal obstruction | 1 week
  measured by acoustical rhinometry and Peak Nasal Inspiratory Flow (PNIF).

CONTACTS AND LOCATIONS:
Overall Officials: Ståle S. Nordgård, MD PhD, Principal Investigator — Aleris/NTNU
Locations (1):
- St Olavs Hospital Trondheim University Hospital, Trondheim, Norway

REFERENCES:
- [Result] Moxness MH, Bugten V, Thorstensen WM, Nordgard S, Bruskeland G. A comparison of minimal cross sectional areas, nasal volumes and peak nasal inspiratory flow between patients with obstructive sleep apnea and healthy controls. Rhinology. 2016 Dec 1;54(4):342-347. doi: 10.4193/Rhino16.085. PMID 27591949